CLINICAL TRIAL: NCT03867734
Title: Aztreonam for Pharyngeal Gonorrhea: A Demonstration Study
Brief Title: Aztreonam for Pharyngeal Gonorrhea
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Lindley Barbee, Assistant Professor, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003878-02
Record Dates: First submitted 2019-03-04; First posted 2019-03-08 (Actual); Results first posted 2022-01-06 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Gonorrhea of Pharynx; Gonorrhea
Keywords: aztreonam; treatment study
MeSH Terms: conditions — Gonorrhea | interventions — Aztreonam

STUDY DESIGN:
Intervention Model Description: Demonstration Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 2g Aztreonam (Experimental): Subjects to receive 2g Aztreonam IM for the treatment of gonorrhea
  Interventions: Drug: Aztreonam

INTERVENTIONS:
Drug: Aztreonam — 2g IM Aztreonam

SUMMARY:
The Centers for Disease Control and Prevention has identified antimicrobial-resistant (AMR) Neisseria gonorrhoeae (NG) as one of the nation's top three urgent AMR threats. Since the advent of antibiotics in the 1930s, NG has developed resistance to every first-line antibiotic. Parenteral third-generation cephalosporins are now the only class of drug with consistent efficacy against NG. New therapies are urgently needed. Although some novel antimicrobials are under development, reevaluating older drugs is another option for quickly identifying additional treatments for gonorrhea. We propose a demonstration study to test a single dose of aztreonam for the treatment of pharyngeal gonorrhea. We chose to focus on pharyngeal gonorrhea because these infections are common, play an important role in fostering gonococcal resistance, and are harder to eradicate than genital infections. Although aztreonam appears to be >98.6% efficacious for anogenital NG, its efficacy at the pharynx may be less. Only 8 cases of pharyngeal gonorrhea have been documented to be treated with aztreonam, but of those, only 5 (62.5%) were cured. The dose used in those studies was 1g of aztreonam. Most antibiotics have a lower efficacy at the pharynx than anogenital sites, which is likely due to drug pharmacokinetics, i.e. difficulty in penetrating pharyngeal tissue. Thus, in the proposed study, we plan to treat 50 subjects with untreated pharyngeal gonorrhea with 2g IM Aztreonam.

Objectives:

The proposed study aims to evaluate the efficacy of a single 2g intramuscular (IM) dose of aztreonam in the treatment of pharyngeal gonorrhea. Secondary objectives include documenting the efficacy stratified by minimal inhibitory concentration (MIC) compared with the previously document area under the curve (AUC) in order to estimate a pharmacodynamic criterion. We will also attempt to determine whether aztreonam monotherapy induces antimicrobial resistance among treatment failures. Lastly, we will evaluate the tolerability of 2g of IM aztreonam. The specific aims are:

1. Determine the proportion of persons whose pharyngeal gonococcal infections are cured with a single dose of 2g aztreonam intramuscularly.
2. Determine the proportion of persons with urethral and/or rectal gonorrhea whose infections are cured with a single dose of 2g aztreonam IM.
3. Evaluate the tolerability of 2g IM of aztreonam .
4. Estimate the best pharmacodynamics criterion (i.e. AUC/MIC ratio) for pharyngeal gonorrhea treated with aztreonam using previously published AUC for 2g aztreonam and NG isolate MIC.
5. Among treatment failures, conduct exploratory analyses comparing pre- and post-treatment MIC for evidence of induced resistance.

Study Design: Prospective cohort

Study Population & Inclusion Criteria:

Persons diagnosed with pharyngeal gonorrhea or gonococcal urethritis who are undergoing pharyngeal gonorrhea testing, who are not yet treated.

Intervention: 2g IM aztreonam x 1

Primary Outcome: Negative gonorrhea culture 4-7 days (+/- 1 day) after treatment

Sample Size: 50 persons

ELIGIBILITY:
Inclusion Criteria:

* Persons diagnosed with pharyngeal gonorrhea or gonococcal urethritis who are undergoing pharyngeal gonorrhea testing, who are not yet treated.

Exclusion Criteria:

* Age less than 16 years
* Receipt of antibiotics in ≤30 days
* Known allergy to aztreonam
* History of renal disease (including diagnosis of solitary kidney, chronic renal insufficiency, renal cell carcinoma etc.)
* Concurrent infection with syphilis or chlamydia
* Pregnancy and/or nursing
* Unable to return for a follow-up visit 4-7 days (+/- 1 day).
* Study team's discretion

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindley Barbee, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- Public Health -- Seattle & King County STD Clinic, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barbee LA, Soge OO, Ocbamichael N, LeClair A, Golden MR. Single-Arm Open-Label Clinical Trial of Two Grams of Aztreonam for the Treatment of Neisseria gonorrhoeae. Antimicrob Agents Chemother. 2020 Dec 16;65(1):e01739-20. doi: 10.1128/AAC.01739-20. Print 2020 Dec 16. PMID 33077658

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 2g Aztreonam
Started | 32
Completed | 30
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | 2g Aztreonam
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 32 (21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 32
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 17
Region of Enrollment [Number; unit: participants]
  United States | 32
HIV co-infection [Count of Participants; unit: Participants] | 3
Sex partner by gender [Number; unit: partners]
  Male | 27
  Female | 0
  Trans/nonbinary | 4
Number of oral sex partners in past 2 months (median range) [Median (Full Range); unit: partners] | 4 [1 to 20]

OUTCOME MEASURES:

1. Primary Outcome: Treatment Efficacy of Pharyngeal Gonorrhea as Defined as the Proportion of Study Participants With Positive Pharyngeal Gonorrhea Culture at of Enrollment Whose Test of Cure Pharyngeal Culture is Negative
Description: Negative Test of Cure (i.e. Pharyngeal Gonorrhea Culture) after Treatment
Time Frame: 4-7 days following treatment
Population: Subjects with pharyngeal culture positive for gonorrhea at enrollment
Measure: Count of Participants; unit: Participants
Groups:
- Pharyngeal Gonorrhea -- Evaluable Population: Subjects who were Pharyngeal Gonorrhea Culture Positive at Enrollment and Received 2g Aztreonam intramuscularly (IM) and Returned for Test of Cure (TOC)
Arm/Group | Pharyngeal Gonorrhea -- Evaluable Population
Number analyzed (Participants) | 6
Participants | 2

2. Secondary Outcome: Efficacy of 2 g Aztreonam for N. Gonorrhoeae at Anogenital Sites
Description: Number of individuals with a negative N. gonorrhoeae culture at an anogenital site at test of cure among those who were N. gonorrhoeae culture positive at the respective anatomic site at the enrollment visit.
Time Frame: Test of Cure 4-7 days following treatment
Measure: Count of Participants; unit: Participants
Groups:
- Efficacy of 2g Aztreonam for Urethral Gonorrhea: Subjects with culture-positive urethral gonorrhea who received 2g Aztreonam IM and returned for TOC
  Aztreonam: 2g IM Aztreonam
- Efficacy of 2g Aztreonam for Rectal Gonorrhea: Subjects with culture-positive gonorrhea of the rectum, treated with 2g Aztreonam and returned for TOC
Arm/Group | Efficacy of 2g Aztreonam for Urethral Gonorrhea | Efficacy of 2g Aztreonam for Rectal Gonorrhea
Number analyzed (Participants) | 9 | 4
Participants | 9 | 3

3. Secondary Outcome: Tolerability of 2g Aztreonam IM
Description: Subjects' self-report of injection related pain on a scale from 0 - 10 where 0 is no pain and 10 is the worst pain ever.
Time Frame: Immediately following injection
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- 2g Aztreonam: All subjects who received 2g Aztreonam IM for the treatment of gonorrhea
  Aztreonam: 2g IM Aztreonam
Arm/Group | 2g Aztreonam
Number analyzed (Participants) | 32
score on a scale | 2 [1 to 3]

4. Secondary Outcome: Side Effects of 2g Aztreonam IM
Description: Subject's report of perceived side effects related to study drug based on responses to standard side effect questionnaire.
Time Frame: assessed immediately following injection and 4-7 days after injection
Population: Of the 30 participants who returned for Test of Cure Visit, 6 reported having a possible side effects between treatment and Test of Cure (4-7 days post injection)
Measure: Count of Participants; unit: Participants
Arm/Group | 2g Aztreonam
Number analyzed (Participants) | 30
Participants
  reported having a HEADACHE | 6
  reported having NAUSEA | 1

ADVERSE EVENTS:
Time Frame: Thirty minutes after injections and then over the following 4 - 6 days or until Test of Cure Visit.
Description: We observed participants for 30 minutes following injection of aztreonam for Type 1 allergic reaction (i.e. IgE mediated-anaphylaxis reactions). A study clinician evaluated participants 4-7 days following aztreonam injection and asked about interim side effects. Aztreonam is usually a very well tolerated. Documented side effects (including, neutropenia, eosinophilia, thrombocytopenia, elevated liver function tests, skin rash, diarrhea, nausea, and vomiting) occur in <2% of cases.
Arm/Group | 2g Aztreonam
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 6/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 2g Aztreonam (N=32)
Headache (Nervous system disorders) | 6
Nausea (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/34/NCT03867734/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/34/NCT03867734/ICF_002.pdf